CLINICAL TRIAL: NCT02181166
Title: Diagnosis and Management of Myofascial Pain Syndrome in Women With Mastectomies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Vânia Tie Koga Ferreira, PT, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1158-7302
Record Dates: First submitted 2014-07-01; First posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer; Myofascial Trigger Point
Keywords: Breast Neoplasms; Mastectomy; Myofascial pain syndromes; Physical Therapy Modalities
MeSH Terms: conditions — Breast Neoplasms; Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- kinesiotherapy + High voltage electrical stimulation (Experimental): Same protocol group kinesiotherapy + high voltage electrial stimulation with two rectangular electrodes (3x5 cm) active silicon-carbon and an electrode rectangular dispersive (10x18cm) aluminum wrapped with a damp felt in water. The active electrodes are positioned in central myofascial trigger point of the upper trapezius muscle after application of water soluble gel. The dispersive electrode was placed in the lumbar region. The following parameters will be use: frequency of 10 Hz, twin pulses of 20μs to 100ms between pulses and the maximum voltage tolerated by voluntary until the motor threshold (visible muscle contraction) to increase every five minutes, totaling 30 minutes of stimulation. The negative polarity will be use.
  Interventions: Other: Kinesiotherapy; Other: High voltage electrical stimulation
- Kinesiotherapy group (Experimental): The volunteer will be subjected to the following protocol: These exercises involve stretching of the cervical, anterior and posterior chain of the upper trunk and active mobilization of the cervical, shoulder movements of flexion, extension, abduction and adduction of the shoulder and upper limb. The exercises lasted 50 minutes, with 10 minutes of walking, and stretching was performed with two repetitions of 20 seconds, and active mobilization exercises of three sets of eight repetitions and final relaxation of 10 minutes were performed.
  Interventions: Other: Kinesiotherapy
- kineshioterapy + isquemic compression (Experimental): The same protocol group kinesiotherapy + ischemic compression in central myofascial trigger point of the upper trapezius muscle. This procedure was performed for 90 seconds.
  Interventions: Other: Kinesiotherapy; Other: Isquemic compression

INTERVENTIONS:
Other: Kinesiotherapy
Other: Isquemic compression
  Arms: kineshioterapy + isquemic compression
Other: High voltage electrical stimulation
  Arms: kinesiotherapy + High voltage electrical stimulation

SUMMARY:
Myofascial pain considerably affects women undergoing treatment for breast cancer, is characterized by the presence of myofascial taut bands and trigger points. This study aims to evaluate the effects of ischemic compression, high-voltage electrical stimulation and rehabilitation of kinesio in women with myofascial pain following treatment of breast cancer. This is a randomized blind controlled study. For this, we invited 60 volunteers undergoing treatment for breast cancer, randomized and allocated into three groups: G1 (cinesioterapia), G2 (ischemic compression cinesioterapia +) and G3 (high voltage electrical stimulation cinesioterapia +). The stance, the plantar pressure distribution and the balance will be assessed by means of photogrammetry and baropodometry respectively. Myofascial trigger points will be assessed with the use of infrared thermography, algometry and numerical rating scale of pain (END). Moreover, the quality of life of the volunteers will be assessed by the Functional Assessment of Cancer Therapy-Breast (FACT-B +4). The volunteers will undergo 10 sessions of treatment, and reassessed at the end of treatment and after thirty days. Normality test is used to verify data distribution and consistent statistical test for proper intra and comparisons between groups, being thus considered two factors in the comparisons, time and group. A significance level of 5% is assumed.

ELIGIBILITY:
Inclusion Criteria:

* mastectomy
* aged between 35 and 70 years
* myofascial trigger point in the upper trapezius muscle

Exclusion Criteria:

* metastasis or recurrence of breast cancer
* bilateral mastectomy
* in physiotherapy treatment
* degenerative diseases of the spine
* use of muscle relaxants or anti-inflammatory analgesics in the last week
* report of fibromyalgia

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-01 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pain | 2 years
  Will be apply the following assessment tools: algometry (evaluates pressure pain threshold), and numerical scale of pain assessment (assesses pain intensity).

SECONDARY OUTCOMES:
Quality of life | 2 years
  Through a Functional Assessment of Cancer Therapy- Breast (FACT B + 4).
Skin Temperature | 2 years
  Through of thermograph will be evaluated skin temperature on myofascial trigger points.
Posture | 2 years
  Through computerized photogrammetry postural assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Vânia Ferreira, PT, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- See also: Related Info — http://www.fmrp.usp.br